CLINICAL TRIAL: NCT02022553
Title: Complex Treatment of Rectal Cancer
Brief Title: Procedure RACHEL in Complex Treatment of Rectal Cancer
Acronym: RACHEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Voronezh N.N. Burdenko State Medical Academy (Other)
Responsible Party: Principal Investigator, Korotkich Nikolay Nikolaevich, M.D., Voronezh N.N. Burdenko State Medical Academy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNKOR2013
Record Dates: First submitted 2013-12-19; First posted 2013-12-30 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer T3-4N0-2M0
Keywords: rectal cancer; RACHEL; oil chemoembolization
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rectal cancer, surgery (Experimental)
  Interventions: Procedure: usual rectal cancer surgery
- rectal cancer, RACHEL, surgery (Active Comparator)
  Interventions: Procedure: RACHEL

INTERVENTIONS:
Procedure: usual rectal cancer surgery
  Arms: rectal cancer, surgery
Procedure: RACHEL
  Other Names: selective endoarterial oil chemoembolisation of upper, middle and lower rectal arteries
  Arms: rectal cancer, RACHEL, surgery

SUMMARY:
AIM OF RESEARCH. The aim of our research is to improve the results of the combined treatment of patients with locally advanced rectal cancer using endovascular methods and reservoir and plastic surgery.

TASKS OF RESEARCH.

1. To assess the immediate and long-term results of combined (chemoradiation and surgical) treatment for locally advanced rectal cancer.
2. To make a comparative evaluation of the results of independent surgical and combined (chemoradiation and surgery) treatment of patients with locally advanced rectal cancer.
3. To examine functional results of surgical treatment with the formation of "neosphincter" and "neorectum" in patients with colorectal cancer..
4. To study features of blood supply to the rectum from the pools of the inferior mesenteric and internal iliac arteries, using the method of selective angiography, in connection with the development of endovascular treatment of rectal cancer.
5. To develop and introduce into clinical practice method of one-stage selective intra-arterial oil chemoembolization of upper, middle and lower rectal arteries in patients with locally advanced rectal cancer, who have a contraindication to preoperative radiotherapy.
6. To assess the immediate and long-term results of combined (endovascular and surgical) treatment for locally advanced rectal cancer.
7. To optimize tactics of combined treatment of locally advanced rectal cancer by developing an algorithm of using chemoradiotherapy and endovascular interventions in the preoperative period.

NOVELTY OF RESEARCH.

1. As a result of research will be designed and implemented a new method of selective intra-arterial chemoembolization in rectal arteries preoperatively in patients with locally advanced rectal cancer.
2. Substantiated high effectiveness of the proposed technique for the removal of colonic obstruction and, as a consequence perform radical surgical treatment of these patients.
3. First developed dosage and concentration of chemotherapeutic agent and embolic agent for safe injection when performing selective intra-arterial chemoembolization of rectal arteries.
4. Developed complex techniques of selective intra-arterial chemoembolization of rectal arteries preoperatively in patients with locally advanced rectal cancer.
5. Will be made a comparative analysis of the postoperative period and the evaluation of the quality of life of operated patients Obtained data will be presented for use in clinical practice. POSSIBLE APPLICATION AREAS. Results of the research designed for use in the treatment process of departments of Coloproctology, oncology, as well as the educational process of higher and secondary medical institutions.

EXPECTED EFFECTIVENESS.

It is expected that the use of this method of treatment of patients with locally advanced rectal cancer in clinical practice will provide pronounced effect:

1. Medical and social - improving the quality of care, preservation of social activity of patients, reducing mortality;
2. Economic - reducing the time of patients' treatment and reducing the number of therapeutic manipulation;
3. Science and Technology - improving of the training level of medicine workers in the treatment of patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rectal cancer T3-4N0-2M0
* complication of bowel obstruction
* No allergy on contrast agent
* Previously not operated about rectal cancer
* Not older than 75 years

Exclusion Criteria:

* Older 75 years
* Previously operated about rectal cancer
* Allergy to contrast agent
* No bowel obstruction
* No rectal cancer
* No locally advanced rectal cancer
* Clinical diagnosis of rectal cancer Tis-4N0-2M1 (generalized rectal cancer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
tumor reduction | 5-10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Voronezh Regional Hospital #1, Voronezh, Voronezh Oblast, Russia